CLINICAL TRIAL: NCT05916872
Title: Combined Effects of Proprioceptive Neuromuscular Facilitation and Electrical Muscle Stimulation on Spasticity and Hand Function in Stroke Patients.
Brief Title: Combined Effects of PNF and Electrical Muscle Stimulation on Spasticity and Hand Function in Stroke Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0211
Record Dates: First submitted 2023-06-14; First posted 2023-06-23 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Stroke; Proprioceptive Disorders; Balance; Distorted
Keywords: Stroke; Proprioceptive Disorders; Balance; Distorted
MeSH Terms: conditions — Stroke; Somatosensory Disorders | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: patients will be allocated to two groups by randomization. Patients in Group A will receive Proprioceptive Neuromuscular Facilitation (contract-relax) technique & EMS patients in Group B will receive conventional therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): patients in this group will receive contract relax exercises along with EMS
  Interventions: Other: experimental group
- control group (Active Comparator): patients in groups B will receive conventional therapy.
  Interventions: Other: control group

INTERVENTIONS:
Other: experimental group — Patients will receive Proprioceptive Neuromuscular Facilitation (contract-relax) technique with EMS
  Arms: experimental group
Other: control group — Patients will receive conventional therapy.
  Arms: control group

SUMMARY:
To determine the combined effects of proprioceptive neuromuscular facilitation and electrical muscle stimulation on spasticity and hand function in stroke patients.

DETAILED DESCRIPTION:
It will be a randomized controlled trial. The stroke patients aged between 30-70 years will be included in this study. Participants will be selected with non-probability convenience sampling technique. Participants will be randomly allocated into two groups by lottery method i.e experimental group and control group. The experimental group will receive proprioceptive neuromuscular technique (contract relax-10 repetition) (5-min) and electrical muscle stimulation(10 min) as 15 min session 3 times a week for four weeks while the control group will receive only conventional therapy. The outcome measure will be calculated by modified barthel index, modified ashworth scale and wolf motor function test.

ELIGIBILITY:
Inclusion Criteria:

* Both ischemic and haemorrhagic stroke patients
* Chronic stroke patients from 6 month to 2years
* Mini Mental Scale Examination (MMSE) more than 25

Exclusion Criteria:

* Transient ischemic attack
* Recurrent stroke
* Stroke patient with comorbidity and cardiac disease
* Myopathies

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Modified Barthel Index: | 9 months
  It is used for assessing the activities of daily living. It is composed of 10 questions that link the degree of independence to daily living activities. Collin et, al; proposed amendment in 1988, in which each domain was scored in one-point increments, ranging from 0 to 2 or 3 for each activity with a maximum score of 20 suggesting functional independence. It is highly reliable and has a good correlation with other disability measures.
Modified Ashworth Scale: | 9 months
  Modified Ashworth Scale:
  It is used to assess the spasticity in patients of stroke or spinal cord injury. Scores range from 0 to 4, where lower scores represent normal muscle tone and higher scores represent spasticity. It is characterized by exaggerated deep tendon reflexes that interfere with muscular activity, gait, movement, or speech. It has excellent validity and reliability.

CONTACTS AND LOCATIONS:
Overall Officials: Zeest Hashmi, MSNMPT, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Fedral, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hankey GJ. The global and regional burden of stroke. Lancet Glob Health. 2013 Nov;1(5):e239-40. doi: 10.1016/S2214-109X(13)70095-0. Epub 2013 Oct 24. No abstract available. PMID 25104481
- [Background] Faghri PD, Rodgers MM, Glaser RM, Bors JG, Ho C, Akuthota P. The effects of functional electrical stimulation on shoulder subluxation, arm function recovery, and shoulder pain in hemiplegic stroke patients. Arch Phys Med Rehabil. 1994 Jan;75(1):73-9. PMID 8291967
- [Background] Rong W, Tong KY, Hu XL, Ho SK. Effects of electromyography-driven robot-aided hand training with neuromuscular electrical stimulation on hand control performance after chronic stroke. Disabil Rehabil Assist Technol. 2015 Mar;10(2):149-59. doi: 10.3109/17483107.2013.873491. Epub 2013 Dec 31. PMID 24377757